CLINICAL TRIAL: NCT04986878
Title: Comparison Between the Analgesic Effects of Single Shot Versus Continuous Adductor Canal Block in Patients Undergoing Total Knee Arthroplasty
Brief Title: Single Shot Versus Continuous Adductor Canal Block in Patients Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Huda Fahmy Mahmoud, PhD, Assistant professor of Anesthesia and Intensive Care, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-10-15
Record Dates: First submitted 2021-06-30; First posted 2021-08-03 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Rheumatism Knee

STUDY DESIGN:
Intervention Model Description: The target population of this study will be patients undergoing primary total knee arthroplasty at Aswan l and Assiut university hospitals
Masking Description: A computer-generated randomization table will be used for patient allocation to one of the two study groups, The SACB group, and the CACB group. Randomization was done in blocks of 10 patients each. Patients' assignments were written in a sealed envelope that was only open after the patient consents to the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single shot adductor canal block (Active Comparator): Following sterile preparation and draping, an ultrasound survey of the medial thigh was performed, halfway between the superior anterior iliac spine and the patella. The superficial femoral artery has been identified beneath the sartorius muscle in a short-axis view, with the vein just inferior and the saphenous nerve just lateral to the artery. A 20 Gauge, 120 mm, non-cuttings tip echogenic needle (SonoPlex STIM, Germany) needle was introduced in-plane, and 2 to 3 mL of LA bolus (0.25 % Bupivacaine) was used to confirm proper needle placement in the adductor canal near the saphenous nerve. Then, a bolus of 20 ml of Bupivacaine 0.25 % was injected through the needle
  Interventions: Procedure: single-shot adductor canal block
- Continuous adductor canal block (Active Comparator): a catheter was secured in place using Tegaderm. The catheters were connected to a pump that infused local anesthetic, 20 mL of 0.25 % bupivacaine, followed by 48 hours of continuous infusion of 0.125 % bupivacaine at 5 mL/h.
  Interventions: Procedure: single-shot adductor canal block

INTERVENTIONS:
Procedure: single-shot adductor canal block — An ultrasound machine (Philips; Model: OTD020, AcBel Polytech Inc., Taiwan) with a 5-10 MHz linear probe was used to perform the adductor canal block immediately postoperatively.
  Other Names: Saphenous nerve block

SUMMARY:
Adductor canal block (ACB) has emerged as an option for postoperative regional analgesia in patients undergoing total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Various approaches to the performance of peripheral nerve blocks for postoperative pain control in patients undergoing TKA have been described in the literature. These approaches include lumbar plexus block, femoral nerve block (FNB), with or without a sciatic nerve block, and most recently the ACB. FNB is a commonly used modality for postoperative analgesia after TKA. It is considered by some as the gold standard or the cornerstone of postoperative analgesia after TKA. However, FNB reduces quadriceps muscle strength essential for mobilization and active contribution in any physical rehabilitation program. Quadriceps weakness places the patients at risk of falling. which may be detrimental to postoperative recovery. The ACB has recently emerged as an appealing alternative to FNB as it is predominately a sensory nerve block of a more distal branch of the femoral nerve ( the saphenous nerve).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary total knee arthroplasty with
* American Society of Anesthesiologists (ASA) physical status I -III,
* mentally competent and able to give consent for enrollment in the study.

Exclusion Criteria:

1. Patient younger than 18 years old or older than 70 years old
2. Allergy to local anesthetics, systemic opioids (fentanyl, morphine, hydromorphone, and any of the drugs included in the multimodal perioperative pain protocol.
3. Revision surgeries were excluded.
4. Impaired kidney functions and patients with coagulopathy were also excluded.
5. Chronic pain syndromes and patients with chronic opioid use defined as the use of regular daily doses of systemic narcotics for the past 6 months prior to the surgery.
6. BMI of 40 or more
7. Pregnancy (positive urine pregnancy test result in Preop area on the morning of surgery)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative pain scores by visual analogue score | 48 hours
  visual analogue score is a straight, vertical 10-cm line with the bottom point representing "no pain" = (0cm) and the top point representing "the worst pain you could ever have" = (10 cm).

SECONDARY OUTCOMES:
time to up and go test (minutes) | 48 hours
  determines how long it takes a person to get out of a chair
six-minute walking test | 48 hours
  calculates the distance that can be walked in 6 minutes
the 30-Second Chair test | 48 hours
  determines how many times a person can rise from a chair and sit down again in 30 seconds while keeping their arms crossed over their chest

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Aswan University Hospital, Aswān
  - Huda Fahmy, Aswān